CLINICAL TRIAL: NCT06096688
Title: Discovering New Targets for Hereditary and Sporadic Colorectal and Endometrial Cancer Risk Reduction
Brief Title: Discovering New Targets for Colorectal and Endometrial Cancer Risk Reduction
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1803019093; U01CA233056 (NIH)
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; Endometrial Cancer; Hereditary Cancer Syndromes
Keywords: personal and family history; genomic/epigenetic; polyps; carcinomas; Hereditary Cancer Syndromes; mucosa; blood serum markers; chemoprevention; registry
MeSH Terms: conditions — Colorectal Neoplasms; Endometrial Neoplasms; Neoplastic Syndromes, Hereditary; Polyps; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — BLOOD COLLECTION. Collection of 3-5 tubes of up to 10 ml each will be performed during standard of care blood draws.
  POLYP/TUMOR COLLECTION DURING PROCEDURE. Removal of polyps and/or tumor tissue will be performed according to standard clinical practices during standard clinical care procedures.
  NORMAL MUCOSA/TISSUE COLLECTION DURING PROCEDURE. Removal of normal mucosa will be performed according to standard clinical practices.
  INCOMPLETELY REMOVED POLYP/TUMOR SAMPLES. Lesions that are not or cannot be completely removed will undergo standard biopsy prior to the acquisition of research biopsies.
  RETROSPECTIVELY COLLECTED SAMPLES. The research team member will coordinate with the pathology team or research laboratory personnel to obtain the tissue and/or samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- FAP without treatment with NSAIDs: Patients with the Hereditary Cancer Syndrome known as Familial Adenomatous Polyposis (FAP) undergoing upper or lower endoscopy/surgery without treatment with NSAIDs
- FAP on treatment with NSAIDs: Patients with the Hereditary Cancer Syndrome known as Familial Adenomatous Polyposis (FAP) undergoing upper or lower endoscopy/surgery on treatment with NSAIDs
- HNPCC without treatment with NSAIDs: Patients with the Hereditary Cancer Syndrome known as Hereditary Non-Polyposis Colorectal Cancer (HNPCC) undergoing lower endoscopy/surgery without treatment with NSAIDs
- HNPCC on treatment with NSAIDs: Patients with the Hereditary Cancer Syndrome known as Hereditary Non-Polyposis Colorectal Cancer (HNPCC) undergoing lower endoscopy/surgery on treatment with NSAIDs
- Other Hereditary Colorectal Cancer Syndromes: Other Hereditary Colorectal Cancer Syndromes undergoing lower endoscopy/surgery
- Average-risk population: Average-risk population undergoing lower endoscopy/surgery in the lower gastrointestinal tract.

SUMMARY:
The primary aim of this study is to collect and store data, tissue, and personal and family histories from patients being screened for colorectal cancer and/or endometrial cancer at NYPH and WCM for routine clinical care and to make these available for future use for molecular and mechanistic studies.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) and endometrial cancer (EC) have a highly heritable component. Approximately 25% of CRC or EC patients have another first or second degree relative who are also affected by CRC or EC, and there are at least 32 known high penetrance CRC/EC germline predisposition genes. The overarching goal of this protocol is to (a) facilitate the discoveries of novel mechanisms in intestinal carcinogenesis and genes inducing genetic predisposition, (b) to help identify new genes and proteins that are amenable to targeted therapy and precision prevention drug intervention and biomarker development in Hereditary Cancer Syndromes, (c) to facilitate understanding and learning about ways of how the immune system can be used to recognize and kill tumor cells that carry mutations. To accomplish these goals, we plan to pursue the following aims:

1. To collect tissue and blood samples for storage, so they can be made available to future research studies and scientist aiming to learn more about the underlying causes of gastrointestinal cancers and endometrial cancers, both in patients with hereditary cancer syndromes and in the general population,
2. To develop organoids from adenocarcinomas, polyps, and normal intestinal mucosa samples in patients with Hereditary Cancer Syndromes and a sporadic cohort as a comparator and control. These organoids will be derived from tissue biopsies of different parts of the intestinal tract, other GI organs, and endometrium in order to perform assessment of drug sensitivity and molecular biology experiments to understand the biology and carcinogenesis of the intestine.

To accomplish these goals, we will obtain normal mucosa, polyp tissue and carcinoma (tumor tissue) arising in the upper gastrointestinal tract (mainly the duodenum, but also other potential locations such as the esophagus, GE junction, stomach, and small bowel), lower gastrointestinal tract (mainly the colorectum), paired normal mucosa samples, endometrial tissue, and blood and as a source of genomic DNA, RNA, and protein.

The biospecimen samples will be collected in the context of standard of care (SOC) endoscopic procedure(s) and/or from pathologic specimens obtained during gastrointestinal (GI) endoscopy procedures and surgery performed at Weill Cornell or New York Presbyterian Hospital, including diagnostic testing, clinic and/or treatment visit and/or from residual blood. These tissue samples and blood samples were collected in the context of routine care and procedures performed at Weill-Cornell and NYPH. Biospecimen samples will also be collected in the context of SOC transvaginal ultrasound, hysteroscopy and endometrium biopsy performed at Weill Cornell or New York Presbyterian Hospital, including diagnostic testing, clinic and/or treatment visit.

Blood samples will be collected at the time blood is taken for clinical care. We will register, collect, process and store frozen blood, frozen normal and diseased tissue and FFPE (formalin fixed paraffin embedded) specimens.

This will be an invaluable annotated hereditary CRC/EC registry and tissue repository that will be available to the Weill Cornell Community upon appropriate approval. Subjects that provide informed consent will agree to collection and storage of clinical data. For the purposes of this project, clinical data includes all data collected for standard clinical purposes (e.g., demographics, medical issues, prognostic data, treatment data, outcomes).

ELIGIBILITY:
The following eligibility criteria must be met as follows:

1. Age ≥ 18 years old.
2. One of the following must be met:

   1. Diagnosis of a Hereditary Cancer Syndrome by positive genetic testing and/or clinical criteria to undergo an endoscopy procedure (esophagoduodenoscopy and/or colonoscopy/flexible sigmoidoscopy), or endometrial screening procedure (transvaginal ultrasound and/or hysteroscopy and/or endometrial biopsy), OR
   2. Individuals coming to Weill-Cornell Medicine/NYPH to undergo an endoscopy procedure, transvaginal ultrasound, or hysteroscopy for average-risk (population-based) recommendation OR
   3. Individuals diagnosed with colorectal cancer or endometrial cancer coming to Weill- Cornell Medicine/NYPH for surgical treatment OR
   4. Individuals coming to Weill-Cornell Medicine/NYPH for care such as, but not limited to, diagnostic testing, clinic and/or treatment visit.
3. Willingness and ability to sign informed consent.
4. Ability to read/understand English, Spanish, and/or simplified Chinese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Presbyterian Hospital (NYPH) and Weill Cornell Medicine (WCM) Gastroenterology and Gynecologic Oncology Patients
Sampling Method: Probability Sample
Enrollment: 1120 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Novel mechanisms and genes inducing genetic predisposition to Hereditary Cancer Syndromes | 7 years
  Discover novel mechanisms in intestinal carcinogenesis and genes inducing genetic predisposition to Hereditary Cancer Syndromes.
New genes and proteins for targeted therapy in Hereditary Cancer Syndromes | 7 years
  Identify new genes and proteins that are amenable to targeted therapy and precision prevention drug intervention and biomarker development in Hereditary Cancer Syndromes.
Understanding and learning about the immune system's ability to recognize and kill tumor cells | 7 years
  To facilitate understanding and learning about ways of how the immune system can be used to recognize and kill tumor cells that carry mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Lipkin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NYP/Weill Cornell Medicine, New York, New York, United States